CLINICAL TRIAL: NCT03703856
Title: Biomarker Predictors of Memantine Sensitivity in Patients With Alzheimer's Disease
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Neal R. Swerdlow, M.D., Ph.D., Principal Investigator, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R01AG059640-01 (NIH)
Record Dates: First submitted 2018-10-09; First posted 2018-10-12 (Actual); Results first posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-07

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's Disease; Alzheimer Disease; Alzheimer; AD; Alzheimer's
MeSH Terms: conditions — Alzheimer Disease | interventions — Memantine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Memantine (Other): EAIP are assessed 210 (PPI) and 345 min (MMN, ASSR) after administration of placebo or memantine (MEM 20 mg po), in a randomized order double-blind design. In this arm subjects are administered MEM 20 mg. Pills look identical so both the subject and research staff are blind to condition.
  Interventions: Drug: Memantine

INTERVENTIONS:
Drug: Memantine — Phase 1 will test the acute effects of memantine (20 mg po) vs. placebo (PBO) on early auditory information processing measures in 32 carefully characterized patients with mild-to-moderate severity AD who are not currently taking AD medications. From this "challenge" test, a set of "early auditory information processing memantine sensitivity" measures will be derived for each patient. In Phase 2, all patients will begin an open-label trial of memantine, titrated to 10 mg bid, with outcome measures collected after 8, 16 and 24 weeks of treatment. Medication adjustments are not restricted, and response heterogeneity is anticipated.

SUMMARY:
The effects of the medication, memantine, on brain functions and the symptoms of Alzheimer's Disease will be tested

DETAILED DESCRIPTION:
Memantine (MEM) is an FDA-approved treatment for Alzheimer's Disease (AD), but its clinical effects vary from person-to-person. We have reported that a "test dose" of MEM significantly enhances early auditory information processing (EAIP) indices of brain function in both healthy adults and psychiatric patients, suggesting that these EAIP measures can be used as "biomarker" evidence that - in a given person - MEM is active within brain circuitry relevant to cognition. This study tests the hypothesis that the EAIP response to a "test dose" of MEM can be used to predict which patients with AD will be most vs. least sensitive to the clinical benefits of this medication over a 24-week trial.

Subjects with mild-to-moderate severity AD who meet criteria for study entry come to UCSD where consenting and a comprehensive screening and diagnostic assessment including a physical exam, EKG, and neuropsychological assessment are conducted. In addition, subjects are assessed on the Alzheimer's Disease Assessment Scale (ADAS-cog), which is the primary clinical outcome measure, and behavioral symptoms documented by the Neuropsychiatric Inventory (NPI-Q) and the Geriatric Depression Scale (GDS), which are secondary assessment measures. Blood is collected in order to assess APOE genotype (rs7412, rs429358) and characterize MEM-sensitive vs. -insensitive patients.

After initial screening, subjects return twice, approximately 7 days apart, for biomarker assessment after challenge with placebo (PBO) or memantine 20 mg po (MEM) in a double-blind, randomized order cross-over design. Subjects are assessed on prepulse inhibition of acoustic startle (PPI), mismatch negativity (MMN) and auditory steady state response (ASSR) as well as AD-relevant cognitive measures via the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS).

Subjects then enter the "treatment phase." MEM is initiated at 5 mg/d and titrated with 5 mg weekly increments. During this time, subjects / caregivers are contacted weekly by study staff to assess adherence. Intervention Week 1 will begin when dosing reaches the full dose of 10 mg bid.

Subjects are reassessed on the primary (ADAS-cog) and secondary (NPI-Q and GDS) outcome measures after 8, 16 and 24 weeks of treatment at the full dose. Subjects are then offered the opportunity to remain at this dose of MEM, or to taper off MEM, under the care of their primary provider.

ELIGIBILITY:
Inclusion:

1. Alzheimer's Disease Research Center-confirmed diagnosis of AD
2. Mini-Mental State Examination (MMSE) score 10-22 OR a Montreal Cognitive Assessment (MOCA) score of 15-24
3. Age 50-83 y
4. Knowledgeable caregiver
5. Ambulatory
6. Medically stable;
7. Audiometric testing (detection < or = to 45 db(A) at 1000 Hz)
8. Informed consent

Exclusion:

1. Active systemic illness (e.g. heart disease, liver failure, renal insufficiency, cancer, HIV, tuberculosis, Hepatitis C)
2. Current psychiatric or neurologic illness other than AD
3. History of vascular disease, myocardial infarction, cerebrovascular accidents, transient ischemic attack, seizure, head injury with loss of consciousness; substance dependence (including alcohol and Opioid)
4. Past treatment with memantine; unable to tolerate acetylcholinesterase inhibitor
5. Investigational drug treatment < 30 d of screening
6. Current meds: amantadine, riluzole, other pro-cognitive medication, opioids
7. Positive urine toxicology for non-prescribed psychoactive substance
8. Actively enrolled in cognitive remediation therapy

Ages: 50 Years to 83 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2025-01-08 (Actual); Study Completion 2025-12-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Neal Swerdlow, M.D., Ph.D., Principal Investigator — UCSD
Locations (1):
- Clinical Teaching Facility (CTF-B102) at UCSD Medical Center, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Enrolled in study
Arm/Group | Memantine
Started | 53
Completed | 30
Not Completed | 23
Not completed — Withdrawal by Subject | 23
Period: Titrated to full dose
Arm/Group | Memantine
Started | 30
Completed | 25
Not Completed | 5
Not completed — Withdrawal by Subject | 5
Period: 8 week assessment
Arm/Group | Memantine
Started | 25
Completed | 25
Not Completed | 0
Period: 16 week assessment
Arm/Group | Memantine
Started | 25
Completed | 24
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: 24 week assessment
Arm/Group | Memantine
Started | 24
Completed | 23
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Includes all subjects consented/enrolled in the study
Arm/Group | Memantine
Number analyzed (Participants) | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.61 (6.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 48
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 42
  More than one race | 0
  Unknown or Not Reported | 6

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Measure in Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-cog) at 8, 16 and 24 Weeks
Description: The Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog) is a tool used to assess the severity of cognitive impairment in individuals with Alzheimer's disease. It includes 11 tasks that evaluate memory, language, and praxis. The total score can range from 0 to 70 with higher scores indicating more severe impairment.
Time Frame: 0, 8, 16, 24 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Memantine
Number analyzed (Participants) | 23
scores on a scale
  Baseline | 19.76 (8.97)
  Week 8 | 19.81 (9.85)
  Week 16 | 19.94 (9.55)
  Week 24 | 20.79 (11.03)
Statistical Analysis 1: Comparison: Memantine; Change in ADAS-Cog score over time; Test type: Superiority; p = 0.68, ANOVA — The threshold for statistical significance was p=0.05

2. Secondary Outcome: Change From Baseline Measure in Neuropsychiatric Inventory-Questionnaire (NPI-Q) at 8, 16 and 24 Weeks
Description: The NPI-Q measures behavioral symptoms in and is a self-administered questionnaire completed by informants about patients for whom they care. Each of the 12 NPI-Q domains contains a survey question that reflects cardinal symptoms of that domain. Symptoms are rated as present or absent, and if they are present the informant rates the severity of the symptom on a 3-point scale from mild to severe. The sum of severity scores across all 12 items ranges from 0 to 36 with higher scores indicate higher severity of symptoms.
Time Frame: 0, 8, 16, 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Memantine
Number analyzed (Participants) | 53
score on a scale
  Baseline | 4.27 (4.05)
  Week 8 | 3.55 (3.36)
  Week 16 | 3.05 (2.38)
  Week 24 | 4.09 (3.57)
Statistical Analysis 1: Comparison: Memantine; Test type: Superiority; p > 0.05, ANOVA — The threshold for statistical significance was p=0.05

3. Other Pre Specified Outcome: Change From Baseline Measure in Geriatric Depression Scale (GDS) at 8, 16 and 24 Weeks
Description: The Geriatric Depression Scale (GDS) is a self-report measure of depression in older adults using a "Yes/No" format. The GDS consists of 30 items with higher scores indicating greater levels or depression. A score of 0-9 is normal, 10-19 is mild depression, and 20-30 is severe depression.
Time Frame: 0, 8, 16, 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Memantine
Number analyzed (Participants) | 53
score on a scale
  Baseline | 6.23 (5.66)
  Week 8 | 6.05 (5.92)
  Week 16 | 6.09 (6.69)
  Week 24 | 6.64 (6.89)
Statistical Analysis 1: Comparison: Memantine; Test type: Superiority; p > 0.05, ANOVA — The threshold for statistical significance is p=0.05

ADVERSE EVENTS:
Time Frame: From enrollment until end of last visit at 24 weeks
Arm/Group | Memantine
All-Cause Mortality (participants affected / at risk) | 0/53
Serious Adverse Events (participants affected / at risk) | 2/53
Other Adverse Events (participants affected / at risk) | 13/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Memantine (N=53)
Abnormal blood test presumed Chronic Lymphocytic Leukemia (Blood and lymphatic system disorders) | 1
Positive prostate biopsy (Reproductive system and breast disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Memantine (N=53)
Dizziness (General disorders) | 3 (3) — Dizziness
Fatigue (General disorders) | 4 (5) — Fatigue
Nausea (Gastrointestinal disorders) | 2 (4) — Nausea
Weight loss (General disorders) | 2 (3) — Weight loss
Constipation (Gastrointestinal disorders) | 2 (2) — Constipation
Tinnitis (Ear and labyrinth disorders) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1) — Fall
Bump in left ear (Ear and labyrinth disorders) | 1 (1) — Bump in left ear
Facial rash (Skin and subcutaneous tissue disorders) | 1 (1) — Facial rash
Foot cramps (Musculoskeletal and connective tissue disorders) | 1 (1) — Foot cramps
Increased EtOH sensitivity (General disorders) | 1 (1) — Increased EtOH sensitivity
Numbness in extremity (Nervous system disorders) | 1 (1) — Numbness in extremity
Positive COVID (Infections and infestations) | 1 (1) — Positive COVID
Visual changes in color perception (Eye disorders) | 1 (1) — Visual changes in color perception
Swelling, forearm (Musculoskeletal and connective tissue disorders) | 1 (1) — Swelling, forearm
Unsteady gait (General disorders) | 1 (1) — Unsteady gait

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-12-05): https://cdn.clinicaltrials.gov/large-docs/56/NCT03703856/Prot_SAP_001.pdf
  • Informed Consent Form (2022-05-02): https://cdn.clinicaltrials.gov/large-docs/56/NCT03703856/ICF_000.pdf